CLINICAL TRIAL: NCT05673122
Title: Socket-Shield Technique With Immediate Implant Placement for Labial Bone Preservation
Brief Title: Socket-Shield Technique With Immediate Implant
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Asrar Moustafa Muftah Althabet, DR, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: socket shield
Record Dates: First submitted 2023-01-03; First posted 2023-01-06 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: Immediate Implants
Keywords: extraction socket; immediate implants; socket shield; labial bone thickness

STUDY DESIGN:
Intervention Model Description: Twenty patients were randomly assigned by specific computer software into two groups either in group (I) or group (II).
  Group I: Ten patients undergo flapless single immediate implant placement surgery with socket shield technique, the implant is in contact with the shield.
  Group II: Ten patients undergo flapless single immediate implant placement surgery with socket shield technique, there was a jumping gap more than 2mm between the shield and the implant, in which the gap was grafted with Xenograft.
Who Masked: Participant
Masking Description: The patients were assigned in two allocated groups using computer randomization "random allocation software" into one of the 2 groups
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Implant intact with shield (Experimental): Ten patients undergo flapless single immediate implant placement surgery with socket shield technique, the implant is in contact with the shield.
  Interventions: Device: Implant(Flotecno)
- Implant not intact with shield (Experimental): Ten patients undergo flapless single immediate implant placement surgery with socket shield technique, there was a jumping gap more than 2mm between the shield and the implant, in which the gap was grafted with Xenograft.
  Interventions: Device: Implant(Flotecno)

INTERVENTIONS:
Device: Implant(Flotecno) — The implants It has a tapered body design and Sandblasting with Large grit that facilitates the osseointergration process.
  made in Italy Flotecno srl via.Turati,38 20121 MILANO (Italia)

SUMMARY:
Primary Objective:

Evaluate of labial plate of bone changes using immediate implant with the socket shield technique in anterior esthetic zone.

Secondary Objective:

Evaluate of soft tissue changes using the immediate implant with socket shield technique in anterior esthetic zone.

DETAILED DESCRIPTION:
Dental implants have become a standard treatment in the replacement of missing teeth. After tooth extraction and implant placement, resorption of buccal bundle bone can pose a significant complication with often very negative cosmetic impacts. Remodeling of the labial bone plate after extraction is a common challenge that affects the final esthetic outcome especially in the esthetic zone.

In addition to, marked bone loss in the horizontal plane and vertical height of the socket wall occurs during the first year after extraction, and one third of this total bone loss occurs during the first three months.

As the buccal aspect of the dental implant has great importance, especially in the aesthetic zone, because the buccal bone is very thin especially in the anterior maxilla and its resorption can result in recession of the soft tissue.

It was suggested that following tooth extraction, the blood vessels in periodontium to the thin bone walls are severed, thereby causing facial bone plate resorption. Thus, it can be assumed that retaining a root may alter the occurrence of facial bone resorption. Many studies showed that the retention of the decoronated root, vital or endodontically treated as root submerge technique, can preserve the alveolar bone.

Other studies also proved that the placement of the implant in contact with retained root surface preserved the buccal bone and led to good emergence profile, Hürzeler et al. (2010) were the first to demonstrate the socket-shield technique in a study on one beagle dog. Were Modification of original technique was done by many researchers by preserving the palatal bone and proximal bone. The promising result of this study shows socket shield technique as a feasible alternative treatment option for thin buccal plate region area and periodontally healthy teeth.

Flapless technique can decrease the amount of bone resorption. Thus, helping in preservation of the inter-dental papilla. Also, it provides less traumatic surgery, decreased operative time, rapid healing and less postoperative complications.

The socket-shield (SS) technique provides a promising treatment adjunct to better manage these risks and preserve the post-extraction tissues in aesthetically challenging cases. The principle is to prepare the root of a tooth indicated for extraction in such a manner that the buccal / facial root section remains in-situ with its physiologic relation to the buccal plate intact.

The socket shield procedure is a novel technique for post extraction implant placement. Several modifications of partial extraction therapy and simultaneous implant placement have been presented since its inception. In this study we discuss the most contemporary step-by-step surgical technique of the socket shield procedure with detailed illustrations and representative cases.

ELIGIBILITY:
Inclusion Criteria:.1. Healthy adlult patient 2. Age from 20-50 years old. 3 Tooth involved in the esthetic zone. 4. Socket Type I. (Elian et al., 2007) 5. Natural teeth adjacent to the involved tooth should be free from periapcial infection.

6. Sufficient hard and soft tissue volume in vertical and buccolingual direction (Levine et al., 2014) 7. Good oral hygiene. 8. Indication for tooth extraction included :( Degidi et al., 2010)

* Non-restorable teeth
* Remaining roots
* Endodontic failures

Exclusion Criteria :1. Presence of acute dento-alveolar infection of involved tooth.

2. Pregnant and breast feeding. 3. Smokers. (Takamiya et al., 2013) 4. Decision impaired individuals (prisoners, handicapped, and mentally retarded) 5. Vertical or Horizontal root fractures on buccal aspect below bone level. 6. External or internal root resorption.

-

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
change of labial bone thickness | baseline at day of surgery and after 6 months
  With the help of CBCT ;Horizontal bone level measurement: Three horizontal lines are drawn 2, 4, and 6 mm apical to implant platform to outer surface of buccal plate of bone. Facial plate of bone is taken as a reference point and is measured baseline (after implant placement and at 6 months follow up).

SECONDARY OUTCOMES:
Pink esthetic score (PES) | baseline presurgery and after 6 months
  Pink esthetic evaluation criteria:
  The Pink Esthetic Score is based on seven variables: mesial papilla, distal papilla, soft-tissue level, soft tissue contour, alveolar process deficiency, soft-tissue color and texture. Each variable was assessed with a 2-1-0 score, with 2 being the best and 0 being the poorest score.
  The mesial and distal papilla were evaluated for completeness, incompleteness or absence. All other variables were assessed by comparison with a reference tooth, i.e., the corresponding tooth (anterior region) or a neighboring tooth (pre-molar region) or evaluate (PES) evaluation before extraction and at six months follow up of involved tooth.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A Hassan, Prof.Dr, Study Chair — Ain Shams University; Asrar M Althabet, MSC, Principal Investigator — Faculty of dentistry Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Nasr City, Egypt

REFERENCES:
- [Background] Abdullah AH, Abdel Gaber HK, Adel-Khattab D. Evaluation of soft tissue and labial plate of bone stability with immediate implant in direct contact versus gap with socket shield: A randomized clinical trial with 1 year follow-up. Clin Implant Dent Relat Res. 2022 Oct;24(5):548-558. doi: 10.1111/cid.13117. Epub 2022 Jun 28. PMID 35763398
- [Background] Degidi M, Daprile G, Piattelli A. Determination of primary stability: a comparison of the surgeon's perception and objective measurements. Int J Oral Maxillofac Implants. 2010 May-Jun;25(3):558-61. PMID 20556255
- [Background] Furhauser R, Florescu D, Benesch T, Haas R, Mailath G, Watzek G. Evaluation of soft tissue around single-tooth implant crowns: the pink esthetic score. Clin Oral Implants Res. 2005 Dec;16(6):639-44. doi: 10.1111/j.1600-0501.2005.01193.x. PMID 16307569
- [Background] Salama M, Ishikawa T, Salama H, Funato A, Garber D. Advantages of the root submergence technique for pontic site development in esthetic implant therapy. Int J Periodontics Restorative Dent. 2007 Dec;27(6):521-7. PMID 18092446
- [Background] Gluckman H, Nagy K, Du Toit J. Prosthetic management of implants placed with the socket-shield technique. J Prosthet Dent. 2019 Apr;121(4):581-585. doi: 10.1016/j.prosdent.2018.06.009. Epub 2018 Dec 13. PMID 30554825
- [Background] Mourya A, Mishra SK, Gaddale R, Chowdhary R. Socket-shield technique for implant placement to stabilize the facial gingival and osseous architecture: A systematic review. J Investig Clin Dent. 2019 Nov;10(4):e12449. doi: 10.1111/jicd.12449. Epub 2019 Aug 21. PMID 31433130
- [Background] Lin X, Gao Y, Ding X, Zheng X. Socket shield technique: A systemic review and meta-analysis. J Prosthodont Res. 2022 Apr 27;66(2):226-235. doi: 10.2186/jpr.JPR_D_20_00262. Epub 2021 Sep 16. PMID 34526435
- [Background] Lang NP, Pun L, Lau KY, Li KY, Wong MC. A systematic review on survival and success rates of implants placed immediately into fresh extraction sockets after at least 1 year. Clin Oral Implants Res. 2012 Feb;23 Suppl 5:39-66. doi: 10.1111/j.1600-0501.2011.02372.x. PMID 22211305
- [Background] Hurzeler MB, Zuhr O, Schupbach P, Rebele SF, Emmanouilidis N, Fickl S. The socket-shield technique: a proof-of-principle report. J Clin Periodontol. 2010 Sep;37(9):855-62. doi: 10.1111/j.1600-051X.2010.01595.x. PMID 20712701
- [Background] Vittorini Orgeas G, Clementini M, De Risi V, de Sanctis M. Surgical techniques for alveolar socket preservation: a systematic review. Int J Oral Maxillofac Implants. 2013 Jul-Aug;28(4):1049-61. doi: 10.11607/jomi.2670. PMID 23869363